CLINICAL TRIAL: NCT00005843
Title: Phase II Trial of R115777 (NSC-702818), an Inhibitor of Farnesyl Protein Transferase, in Patients With Previously Untreated Metastatic Pancreatic Adenocarcinoma
Brief Title: R115777 in Treating Patients Who Have Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02335; FCCC-00005; NCI-45; CDR0000067859 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-06-02; First posted 2004-03-05 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2007-04

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — tipifarnib

ARMS (1):
- Arm I (Experimental): Patients receive oral R115777 twice daily for 21 consecutive days. Treatment continues every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tipifarnib

INTERVENTIONS:
Drug: tipifarnib

SUMMARY:
Phase II trial to study the effectiveness of R115777 in treating patients who have metastatic pancreatic cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the safety and effectiveness of R115777 in patients with metastatic pancreatic cancer.

II. Determine the response rate, time to progression, and 6 month survival rate of these patients with this treatment regimen.

III. Assess the pharmacokinetics of this treatment regimen in this patient population.

OUTLINE: This is a multicenter study.

Patients receive oral R115777 twice daily for 21 consecutive days. Treatment continues every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the pancreas
* Measurable metastatic disease No prior treatment for metastatic disease except immunotherapy (e.g., antibodies, vaccines, cytokines)

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: ECOG 0-2
* WBC at least 4,000/mm3 OR granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Bilirubin no greater than 2.0 mg/dL
* SGOT/SGPT no greater than 2 times normal
* Creatinine no greater than 2.0 mg/dL OR creatinine clearance at least 50 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months after the study
* No concurrent illness or active infection which would preclude study
* No prior malignancy allowed unless disease free for the time period considered appropriate for cure of the specific cancer
* No history of allergies to imidazole compounds (e.g., fluconazole, ketoconazole, miconazole, itraconazole, clotrimazole)

PRIOR CONCURRENT THERAPY:

* No prophylactic filgrastim (G-CSF), sargramostim (GM-CSF), or thrombopoietin
* Primary neoadjuvant or adjuvant chemotherapy allowed at least 6 months prior to detection of metastatic disease
* Primary radiotherapy allowed at least 6 months prior to detection of metastatic disease
* No concurrent use of proton pump inhibitors (e.g., omeprazole)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2000-05; Primary Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal J. Meropol, MD, Study Chair — Fox Chase Cancer Center
Locations (2):
- United States (2):
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Texas - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Cohen SJ, Ho L, Ranganathan S, Abbruzzese JL, Alpaugh RK, Beard M, Lewis NL, McLaughlin S, Rogatko A, Perez-Ruixo JJ, Thistle AM, Verhaeghe T, Wang H, Weiner LM, Wright JJ, Hudes GR, Meropol NJ. Phase II and pharmacodynamic study of the farnesyltransferase inhibitor R115777 as initial therapy in patients with metastatic pancreatic adenocarcinoma. J Clin Oncol. 2003 Apr 1;21(7):1301-6. doi: 10.1200/JCO.2003.08.040. PMID 12663718